CLINICAL TRIAL: NCT01832064
Title: Development of a Mailed Chronic Disease Self-Management Program
Brief Title: Active Living Tool Kit for Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 26610
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Diseases
Keywords: chronic disease; patient education; self management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mailed Chronic Disease Self-Management (Experimental): Mailed Chronic Disease Self-Management Program: self management information and self assessment
  Interventions: Behavioral: Mailed Chronic Disease Self-Management Program

INTERVENTIONS:
Behavioral: Mailed Chronic Disease Self-Management Program — materials are mailed to participants

SUMMARY:
The development and pilot testing of a self-management program that would be delivered in a one time mailing.

DETAILED DESCRIPTION:
The mailing will consist of (1) A self-test that will help users know how he or she can best use the materials and where to start; (2) A copy of the 2012 Living Healthy Life with Chronic Conditions book. If people are visually impaired or have low literacy an audio CD of the book will be available in place of the print copy; (3)An exercise CD with flexibility and strengthening exercises at three different levels of intensity, designed for people with chronic conditions; (4) A relaxation CD with three different relaxation exercises; and (5) In addition, there will be tip sheets, one for each major tool such as managing pain, managing sleep, etc. It is expected that there will be 10-20 tip sheets in total.

The key content of the self-test and the tip sheets will be developed surveying master trainers of the existing small-group Chronic Disease Self Management Program (100 active trainers) and asking about 500 additional trainers to rank importance of key content items generated in initial survey. Pilot testing of the program will be by 250 people with chronic diseases. Participants will be surveyed by mailed questionnaires at baseline and six-months. A subgroup with diabetes (estimated 25-30%) will be asked to submit hemoglobin A1C blood test kits at baseline and six months.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic health condition
* 18 years of age
* Literate in English
* (for the blood test subset): have type 2 diabetes

Exclusion Criteria:

* Taken the small group or online Chronic Disease Self Management Program or related programs
* under 18
* active cancer treatment
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Health Status (symptoms, activity limitation) | six months

SECONDARY OUTCOMES:
Metabolic control (HbA1c) | six months
  For subset of participants with type 2 diabetics
health behavior (exercise, communication with physician) | six months
Health care utilization | six months
  MD, emergency, hospital times and total nights

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lorig, DPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicien, Stanford, California, United States